CLINICAL TRIAL: NCT05914909
Title: A Phase 1, Randomised, Placebo-controlled Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of 10 mg/kg AD-214 When Administered Intravenously to Healthy Volunteers and Patients With Interstitial Lung Disease or Chronic Kidney Disease
Brief Title: Safety, Tolerability, PK and PD Study of AD-214 Administered to Healthy Volunteers and Patients With Interstitial Lung Disease or Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AdAlta Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1AD-AD-214-2301
Record Dates: First submitted 2023-05-28; First posted 2023-06-22 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Interstitial Lung Disease; Chronic Kidney Diseases
MeSH Terms: conditions — Lung Diseases, Interstitial; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: AD-214 in Healthy Volunteers (Experimental)
  Interventions: Biological: AD-214
- Part A: Placebo in Healthy Volunteers (Placebo Comparator)
  Interventions: Other: Placebo
- Part B: AD-214 in patients with ILD or CKD (Experimental)
  Interventions: Biological: AD-214
- Part B: Placebo in patients with ILD or CKD (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AD-214 — AD-214 is a recombinant Fc-fusion protein that selectively binds to CXCR4 to antagonise the SDF-1/CXCR4 axis.
  Arms: Part A: AD-214 in Healthy Volunteers; Part B: AD-214 in patients with ILD or CKD
Other: Placebo — Placebo
  Arms: Part A: Placebo in Healthy Volunteers; Part B: Placebo in patients with ILD or CKD

SUMMARY:
This is a Phase I, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of a 10 mg/kg dose of AD-214 when administered to healthy volunteers (HVs) (Part A) or patients with interstitial lung disease (ILD) or chronic kidney disease (CKD) (Part B). The study will be performed in Australia at up to two clinical sites.

ELIGIBILITY:
Inclusion Criteria:

* All Study Parts:

  1. Male or female aged ≥ 18 to ≤ 65 years of age at the time of consent.
  2. Provision of signed informed consent prior to study entry and agreement to adhere to all study protocol requirements.
  3. Agreement to adhere to the current state and national advice regarding minimising exposure to corona virus disease from the first screening visit until the EoS visit.
  4. Maximum weight of 100.00 kg and BMI > 18.0 and < 30.0 kg/m2 (inclusive) at the time of consent. Participants must also be < 100.00 kg at Day -1.
  5. Normal vital signs after ≥ 5 minutes resting supine position:

     * > 90 mmHg and <160 mmHg SBP
     * 50 mmHg and < 95 mmHg DBP
     * > 45 bpm and < 101 bpm HR
     * Body temperature >35.5oC and ≤37.6°C
  6. Ability and willingness to attend the necessary visits to the CRU.
  7. Have established use of highly effective, double barrier contraception (both partners) prior to screening, during the study AND for 90 days following completion of dosing as specified below in this criterion.

     Double barrier contraception is defined as a condom AND 1 other form of the following:
     * Hormonal and non-hormonal forms of contraception (including oral, depot or injectable)
     * IUD/IUS
     * Sterilised male partner. Rhythm methods will not be considered as highly effective methods of birth control.

     Participant abstinence from heterosexual sexual activity, if their usual and preferred lifestyle, for the duration of the study and for 90 days after the last dose of AD-214 is acceptable.

     Participants who are in a same sex relationship will not require contraception unless they enter into a heterosexual relationship.

     Female participants and female partners of male participants must use double barrier contraception including condom from start of study and for 90 days after last dose of AD-214.
  8. Male participants must refrain from sperm donation and female participants must refrain from ova donation from the first dose of AD-214 and for 90 days after last dose of AD-214.
  9. WOCBP must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1. Females not of childbearing potential must be surgically sterile or post-menopausal (defined as cessation of regular menstrual periods for at least 12 months), confirmed by FSH level at Screening.
  10. Must not regularly consume more than 10 standard alcoholic drinks in a week and more than 4 standard alcoholic drinks in any one day for the duration of the study, AND must for the duration of the study agree to:

      * abstain from alcohol intake from 48 hours before each study drug administration through to discharge from the CRU AND
      * abstain from alcohol intake from 24 hours before each outpatient study visit.
  11. Must not be a regular smoker of > 5 cigarettes/e-cigarettes/cigars/pipes a day AND must, for the duration of the study, agree to:

      * smoke no more than 5 cigarettes/ e-cigarettes/cigars/pipes in any 1 day from 48 hours before first study drug administration until the EoS visit
      * abstain from smoking 24 hours before each study drug administration through to discharge from the CRU
      * abstain from smoking from 24 hours before each outpatient study visit.

      Part A: HVs only
  12. Must be in good general health, in the opinion of the Investigator, with no significant medical history, have no clinically significant abnormalities on physical examination at Screening, and/or before administration of the initial dose of study drug.
  13. Must have clinical laboratory values within normal range in the opinion of the Investigator. Repeat screening may be permitted if out of range values are deemed NCS by the Investigator. Exercise induced elevated creatinine kinase levels may be permitted if out of range values are deemed NCS by the Investigator.

      Part B: Patients with ILD or CKD
  14. Clinical and radiological features that are consistent with an established diagnosis of any of the following diseases in which high expression of CXCR4 has been implicated ;

      * CKD due to LN, DN, and FSGS OR
      * IPF OR fibrotic ILD associated with any of the following: CVD, Fibrotic non-specific interstitial pneumonia (fNSIP), Chronic fibrosing hypersensitivity pneumonitis (cHP)
  15. Must be on a stable regimen of systemic medications for their ILD or CKD and expected to continue on this regimen until completion of the final EoS visit.

      Patients with ILD:
  16. Most recent HRCT image (taken within 12 months of Screening) showing either UIP pattern as per current ATS/ ERS/ JRS/ALAT guidelines in IPF patients, OR, for patients with fibrotic ILD, a > 10% extent of fibrosing lung disease.
  17. Predicted FVC ≥ 50% on PFTs conducted within 3 months of Screening.
  18. Predicted haemoglobin-corrected DLCO ≥ 25% in PFTs conducted within 6 months of Screening.

      Patients with CKD:
  19. Estimated glomerular filtration rate greater than or equal to 30 mL/min/1.73 m2
  20. Proteinuria ≥ 1 based on absolute amount in grams per day (g/d) as measured in 1 complete and valid 24-hour urine collection during Screening.

Exclusion Criteria:

* All Study Parts:

  1. Previously received AD-214
  2. Received any IMP within 30 days or 5 half-lives prior to Screening, whichever is longer.
  3. Received an investigational vaccine, recombinant protein or monoclonal antibody within 6 months, a live attenuated registered vaccine within 60 days, or a registered vaccine within 30 days prior to the first dose of the IP.
  4. Received blood or blood products within 1 month prior to Screening.
  5. Blood donation or significant blood loss (> 280 mL) within 60 days prior to the first dose of the IP.
  6. Plasma donation within 7 days prior to the first dose of the IP.
  7. A bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with blood draws.
  8. Unable to provide a blood sample without undue trauma or distress or inadequate venous access.
  9. Recent (less than 6 weeks) significant wound (in the opinion of the PI), or presence of an ongoing non-healing skin wound on Day -1.
  10. Positive test for HIV, HBsAg, or anti-HCV at Screening.
  11. A psychiatric condition that precludes compliance with the protocol in the opinion of the Investigator; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to Screening, a history of suicide plan.
  12. Clinical signs of active infection and/or a temperature of > 37.7°C at the time of Screening. Study entry may be deferred at the discretion of the PI.
  13. Fever in the past 7 days within Screening or Day 1 AND symptoms reflective of an active respiratory tract infection (in the opinion of the Investigator).
  14. QTcF > 450 msec for females and > 470 msec for males, or QTcF > 480 msec in participants with Bundle Branch Block.
  15. Active malignancy and/or history of malignancy in the past 5 years, with the exception of non-melanoma skin cancer, or low grade cervical intraepithelial neoplasia.
  16. A history of severe allergic, anaphylactic, or other hypersensitive reactions to AD-214 excipients, a history of drug or other allergy including severe allergic reaction that in the opinion of the Investigator or Sponsor MM contraindicates their participation.
  17. Surgery within the past 3 months prior to the first study drug administration determined by the PI to be clinically relevant.
  18. History or presence of alcohol abuse (defined as an average weekly intake of > 10 units. One unit is equivalent to 10 g of alcohol and the following can be used as a guide: a half-pint [~240 mL] of beer, 1 glass [125 mL] of wine or 1 [30 mL] measure of spirits) or drug abuse (including recreational marijuana use) within the 2 years prior to the first study drug administration, and unwillingness to be totally abstinent during the dosing period.
  19. Positive alcohol breath test or urine drugs of abuse screen at Screening or Day -1
  20. Inability to adhere to smoking and alcohol restrictions for the duration of the study.
  21. Pregnant or lactating.

      Part A: HVs:
  22. Any clinically significant abnormality at Screening determined by medical history, physical examination, biochemistry, haematology, coagulation, urinalysis, and 12-lead ECG.
  23. History of recurrent infections, with the exception of urinary tract infections.
  24. Serious (as per the discretion of the PI or Investigator) local infection or systemic infection requiring antibiotic or anti-viral treatment within 3 months from Screening.
  25. Extensive chronic obstructive pulmonary disease including emphysema and chronic bronchitis as judged by the PI or Investigator.
  26. A history of or current chronic medical condition (eg, hypertension, asthma, diabetes, or cardiac disease) or any other medical, social, or psychiatric condition, significant co-morbidities, or any finding during Screening, which in the Investigator's opinion may interfere with the study objectives, may put the participant at risk, or may make the participant unsuitable for participation in the study.
  27. Use of any prescription or over the counter medication (with the exception of paracetamol and contraceptives) within 7 days of first study drug administration.
  28. Any acute illness within 30 days prior to Day 1.

      Part B:

      All Patients
  29. Alanine aminotransferase (ALT) > 2 × ULN and total bilirubin > 1.5 × ULN.
  30. Use of anticoagulants or antiplatelet agents (excluding aspirin).
  31. Severe/significant arterial hypertension, heart failure or coronary heart disease.
  32. Significant hypoxia, requiring > 2 L/min oxygen chronically to maintain a resting oxygen saturation > 89%.

      Patients with ILD
  33. Poor exercise tolerance with 6MWD < 150 metres.
  34. Extensive emphysema on HRCT as defined by being greater in extent than the accompanying fibrotic lung disease.
  35. Evidence of physiologically significant obstructive airways disease as evident from

      * FEV1/FVC ratio < 0.7 OR
      * Bronchodilator response defined by an increase of ≥ 12% and an increase of ≥ 200 mL in the FEV1 after bronchodilator
  36. Other explanation for lung fibrosis, including but not limited to radiation, sarcoidosis, bronchiolitis obliterans organising pneumonia, HIV, viral hepatitis.

      Patients with CKD
  37. Post-transplant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events that are related to treatment in healthy volunteers [Safety and Tolerability] | 141 days
  Safety and Tolerability as assessed by the number of adverse events that are related to treatment versus placebo
Incidence of adverse events that are related to treatment in patients with ILD or CKD [Safety and Tolerability] | 57 days
  Safety and Tolerability as assessed by the number of adverse events that are related to treatment versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Emir Redzepagic, Dr, Principal Investigator — CMAX Clinical Research Pty Ltd
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No